CLINICAL TRIAL: NCT02039050
Title: Proof of Concept Evaluation of Drug-Device Interaction With Aclidinium Bromide Via Genuair® and Tiotropium Bromide Via HandiHaler® in COPD Using Impulse Oscillometry
Brief Title: Evaluation of Long-Acting Muscarinic Antagonists in COPD
Acronym: MAN04
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: Almirall Limited (Unknown)
Responsible Party: Principal Investigator, Brian J Lipworth, Professor of Allergy and Pulmonology, University of Dundee
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2013RC09
Record Dates: First submitted 2014-01-15; First posted 2014-01-17 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary Disease, Chronic Obstructive; Long-acting muscarinic antagonists; Impulse oscillometry
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; aclidinium bromide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tiotropium (Active Comparator): Participants receive tiotropium for 2 to 3 weeks.Participants then enter a washout period and after the washout period receive the alternative treatment arm.
  Interventions: Drug: Tiotropium
- Aclidinium (Experimental): Participants receive tiotropium for 2 to 3 weeks.Participants then enter a washout period and after the washout period receive the alternative treatment arm.
  Interventions: Drug: Aclidinium

INTERVENTIONS:
Drug: Tiotropium
  Arms: Tiotropium
Drug: Aclidinium
  Arms: Aclidinium

SUMMARY:
In chronic obstructive pulmonary disease (COPD), the airways of the lungs are narrowed or blocked. Bronchodilators are drugs usually delivered through inhalers which help open up the airways. Tiotropium is a type of bronchodilator drug known as a long-acting muscarinic antagonist (LAMA). For a long time tiotropium was the only available LAMA. More recently, a new LAMA called aclidinium has been approved for use in COPD. There are potentially important differences between these two medications that might have an impact on the treatment of COPD patients.

In this study we aim to compare the effects of tiotropium and aclidinium in people with COPD. The main comparison will be done using a very sensitive breathing test called impulse oscillometry

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers aged 40-80 years with moderate to severe COPD (GOLD Stage 2, 3).
* On inhaled corticosteroids / long-acting beta agonists
* FEV1 30-80% predicted and FEV1/FVC <70%.
* Smoking history ≥10 pack-years.
* Ability to give informed consent
* Agreement for their General Practitioner to be made aware of study participation and to receive feedback as relevant to the participant's well being

Exclusion Criteria:

* Other respiratory diseases such as asthma, bronchiectasis or allergic bronchopulmonary aspergillosis
* A COPD exacerbation or respiratory tract infection requiring systemic steroids and/or antibiotics within 1 month of the study commencement (3 months if hospitalisation has been required)
* Any clinically significant medical condition that may endanger the health or safety of the participant
* Known or suspected sensitivity to/intolerance of investigational medicinal product
* Patients with prostatic hyperplasia, bladder outflow obstruction or glaucoma
* Pregnancy or lactation
* Unable to comply with the procedures of the protocol

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in trough R5 from baseline after chronic dosing | 4 to 6 weeks

SECONDARY OUTCOMES:
Remaining impulse oscillometry (IOS) variables (R20,R5-R20,X5,AX,RF) | 4 to 6 weeks
Spirometry (FEV1, FEF25-75, FVC) | 4 to 6 weeks
Relaxed VC (RVC) with RVC to FVC ratio | 4 to 6 weeks
Six-minute walk test (includes oxygen saturation measurements and Borg dyspnoea score) | 4 to 6 weeks
Domiciliary PIKO-6 measurements for FEV1 and FEV6 | 4 to 6 weeks
St. George's Respiratory Questionnaire (SGRQ) | 4 to 6 weeks
Baseline Dyspnea Index-Transition Dyspnea Index (BDI-TDI) | 4 to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Brina Lipworth, MD, Principal Investigator — University of Dundee; Arvind Deva Manoharan, MBChB, Principal Investigator — University of Dundee
Locations (1):
- Asthma and Allergy Research Group, University of Dundee, Dundee, United Kingdom

REFERENCES:
- [Result] Manoharan A, Morrison AE, Lipworth BJ. Effects of Adding Tiotropium or Aclidinium as Triple Therapy Using Impulse Oscillometry in COPD. Lung. 2016 Apr;194(2):259-66. doi: 10.1007/s00408-015-9839-y. Epub 2016 Jan 13. PMID 26758884